CLINICAL TRIAL: NCT00196599
Title: Pilot Study on Efficacy and Safety of a Once Daily FTC, ddI, Efavirenz Combination in Antiretroviral Naive HIV Infected Adults. ANRS 091 MONTANA
Brief Title: Pilot Study on Once Daily FTC, ddI, Efavirenz Combination in Antiretroviral Naive HIV Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Triangle Pharmaceuticals (Industry); Gilead Sciences (Industry); Bristol-Myers Squibb (Industry); Dupont Applied Biosciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 091 MONTANA
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections; Antiretroviral Naive
Keywords: HIV infections; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Racivir; Pharmaceutical Preparations; Didanosine; efavirenz

INTERVENTIONS:
Drug: emtricitabine, FTC (drug)
Drug: didanosine, ddI (drug)
Drug: efavirenz (drug)

SUMMARY:
In 1999, when initiating antiretroviral treatment in HIV infected adults, a triple combination with protease inhibitor is recommended. Such therapy induces side effects and the number of pills may reduce therapy adherence. The aim of this study is to evaluate the efficacy and the safety of a once daily FTC, ddI, efavirenz combination, in HIV patients with CD4 cell count over 100/mm3, antiretroviral naive.

DETAILED DESCRIPTION:
In 1999, when initiating antiretroviral treatment in HIV infected adults, a triple combination with protease inhibitor is recommended. Side effects of this products and the number of pills may induce a lower adherence, and thus a lower efficacy. 40 patients with a CD4 count over 100/mm3, a HIV RNA over 5,000 copies/ml and antiretroviral naive, take the once daily combination of FTC, ddI, efavirenz during 24 weeks. The primary end-point is the viral success maintained from 12 weeks until 24 weeks. Secondary end-point is the adherence to the association and safety.

The trial is prolonged during a total of 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Antiretroviral naive
* CD4 cell count over 100/mm3
* Plasma HIV RNA load over 5,000 copies/mL
* Signed written informed consent

Exclusion Criteria:

* Hepatitis B infection
* Pregnancy
* Alcool abuse
* Acute infection, past neurological or pancreatic disease, biological abnormalities
* Chemotherapy or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39
Dates: Start 1999-02; Study Completion 2004-09

PRIMARY OUTCOMES:
Virological success

SECONDARY OUTCOMES:
Treatment adherence
CD4 cell count
Safety
Progression of HIV infection
Pharmacokinetics criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Molina, MD, PhD, Principal Investigator — Service de Maladies Infectieuses, Hôpital Saint-Louis, Paris, 75475, France; Genevieve Chene, MD, PhD, Study Director — INSERM unité 593, Bordeaux, France

REFERENCES:
- [Result] Molina JM, Ferchal F, Rancinan C, Raffi F, Rozenbaum W, Sereni D, Morlat P, Journot V, Decazes JM, Chene G. Once-daily combination therapy with emtricitabine, didanosine, and efavirenz in human immunodeficiency virus-infected patients. J Infect Dis. 2000 Aug;182(2):599-602. doi: 10.1086/315711. Epub 2000 Jul 13. PMID 10915095
- [Result] Molina JM, Peytavin G, Perusat S, Lascoux-Combes C, Sereni D, Rozenbaum W, Chene G. Pharmacokinetics of emtricitabine, didanosine and efavirenz administered once-daily for the treatment of HIV-infected adults (pharmacokinetic substudy of the ANRS 091 trial). HIV Med. 2004 Mar;5(2):99-104. doi: 10.1111/j.1468-1293.2004.00194.x. PMID 15012649